CLINICAL TRIAL: NCT01244191
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of ARQ197 Plus Erlotinib Versus Placebo Plus Erlotinib in Previously Treated Subjects With Locally Advanced or Metastatic, Non-Squamous, Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Tivantinib Plus Erlotinib Versus Placebo Plus Erlotinib for the Treatment of Non-squamous, Non-small-cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision due to the protocol-defined stopping boundary for futility was met based on the interim OS data.
Sponsor: Daiichi Sankyo (Industry)
Collaborators: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARQ197-A-U302; 2010-022365-10 (EudraCT Number)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2020-10-30 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Non Squamous, Non-small-cell Lung Cancer
Keywords: Non squamous, non-small-cell lung cancer; Epidermal growth factor receptor; c-Met inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ARQ 197; Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tivantinib and erlotinib (Experimental): Tivantinib 720 mg daily (360 mg twice a day) in combination with 150 mg of erlotinib, given once a day
  Interventions: Drug: Tivantinib; Drug: Erlotinib
- Placebo and erlotinib (Active Comparator): Tivantinib placebo given twice a day in combination with 150 mg of erlotinib, given once a day
  Interventions: Drug: Placebo; Drug: Erlotinib

INTERVENTIONS:
Drug: Tivantinib — Tivantinib 720 mg daily as 3 x 120 mg oral tablets given twice a day
  Other Names: ARQ197
  Arms: Tivantinib and erlotinib
Drug: Placebo — Tivantinib Placebo tablets given twice a day
  Other Names: No drug
  Arms: Placebo and erlotinib
Drug: Erlotinib — Erlotinib 150 mg oral tablets, given once a day

SUMMARY:
This study is to determine if the combination regimen of tivantinib with erlotinib will improve overall survival relative to erlotinib alone in subjects with locally advanced or metastatic non-squamous, non-small cell lung cancer who have received 1 or 2 prior systemic anti-cancer therapies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed surgically unresectable locally advanced or metastatic (stage IIIB/IV) non-squamous non-small-cell lung cancer.
* Measurable disease and documented disease progression following last prior therapy according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, Version 1.1.
* Have received one or two prior lines of systemic anti-cancer therapy therapy for advanced or metastatic disease, one of which must be a platinum-doublet therapy. Patients who received only adjuvant treatment will be eligible only if disease progression occurred <6 months after completion of adjuvant therapy. Prior maintenance therapy is allowed and will be considered as the same line of therapy when continued without discontinuation after initiation of a treatment regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Resolution of any toxic effects of prior therapy (including radiotherapy) according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0, Grade ≤1 (with the exception of alopecia and ≤grade 2 neuropathy). Subject must have recovered from significant surgery-related complications.
* Demonstrate adequate bone marrow, liver, and renal functions, defined as:
* ALT, AST, and alkaline phosphatase ≤ 2.5 × upper limit of normal (ULN) in subjects with no liver metastasis and ≤5.0 x ULN in subjects with liver metastasis.
* Total bilirubin ≤ 1.5 × ULN (≤ 4 × ULN total and ≤1.5 × ULN direct bilirubin is acceptable for subjects with Gilbert's syndrome).
* ANC ≥1.5 × 10^9/L.
* Platelet count ≥100 × 10^9/L.
* Hemoglobin ≥9.0 g/dL (transfusion and/or growth factor support allowed).
* Serum creatinine ≤1.5 × ULN or creatinine clearance ≥ 60 mL/min.
* Archival and/or fresh biopsy tissue sample must be available for biomarker determination. The status of the following biomarkers will be collected in this study: EGFR and KRAS mutation status prior to randomization, and MET status post randomization
* If of child-bearing/reproductive potential (female or male), must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received
* If female and of childbearing potential, must have a negative result of a pregnancy test (serum or urine) within 72 hours prior to initiating study treatment.
* Must have signed and dated an approved Informed Consent Form (Including HIPAA authorization, if applicable) before performance of any study-specific procedures or tests. Subjects must be fully informed about their illness and the investigational nature of the study protocol (including forseeable risks and possible side effects)

Exclusion Criteria:

* Prior therapy with an EGFR inhibitor and/or ARQ 197 (or other known c-MET inhibitor).
* Receipt of any systemic anti-tumor treatment for NSCLC within 3 weeks prior to randomization.
* Receipt of palliative radiotherapy within 2 weeks or radiotherapy for curative intent of target lesions within 3 weeks prior to randomization. Lesions subjected to radiotherapy within 3 weeks prior to randomization may not be used as target lesions.
* Major surgical procedure within 3 weeks prior to randomization.
* History of cardiac disease:

Congestive heart failure defined as Class II to IV per New York Heart Association classification; active coronary artery disease; previously diagnosed symptomatic bradycardia (subjects with asymptomatic bradycardia and heart rate above 50 bpm are allowed) or other cardiac arrhythmia defined as ≥Grade 2 according to NCI CTCAE, version 4.0, or uncontrolled hypertension; myocardial infarction that occurred within 6 months prior to study entry (myocardial infarction that occurred > 6 months prior to study entry is permitted).

* Clinically unstable central nervous system (CNS) metastasis (to be enrolled in the study, subjects must have confirmation of stable disease by MRI or computed tomography (CT) scan within 4 weeks of randomization and have CNS metastases well controlled by steroids, anti-epileptics or other symptom-relieving medications).
* Need to breastfeed a child during or within 12 weeks of completing the study.
* Significant gastrointestinal disorder that, in the opinion of the investigator, could interfere with absorption of ARQ 197 and/or erlotinib (eg, Crohn's disease, small or large bowel resection, malabsorption syndrome).
* Inability or unwillingness to swallow the complete doses of ARQ 197 or erlotinib.
* Any known contraindication to treatment with, including hypersensitivity to, ARQ 197 or erlotinib.
* History of malignancy other than NSCLC within the 5 years prior to randomization, with the exceptions of adequately treated intraepithelial carcinoma of the cervix uteri; prostate carcinoma with a prostate-specific antigen value <0.2 ng/mL; or basal or squamous-cell carcinoma of the skin.
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Any other significant co-morbid condition that, in opinion of the investigator, would impair study participation or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1048 (Actual)
Dates: Start 2011-01-11 (Actual); Primary Completion 2012-12-15 (Actual); Study Completion 2012-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (257):
- United States (88):
  - Tucson, Arizona
  - Los Angeles, California
  - Oxnard, California
  - Rancho Mirage, California
  - Santa Monica, California
  - Aurora, Colorado
  - Boulder, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Lakewood, Colorado
  - Littleton, Colorado
  - Lone Tree, Colorado
  - Longmont, Colorado
  - Parker, Colorado
  - Thornton, Colorado
  - Newark, Delaware
  - Fort Myers, Florida
  - Miami Beach, Florida
  - Pensacola, Florida
  - Atlanta, Georgia
  - Austell, Georgia
  - Carrollton, Georgia
  - Cartersville, Georgia
  - Douglasville, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Carmel, Indiana
  - Fishers, Indiana
  - Goshen, Indiana
  - Greenfield, Indiana
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Towson, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Grand Island, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - East Orange, New Jersey
  - Albuquerque, New Mexico
  - Buffalo, New York
  - Goshen, New York
  - Latham, New York
  - New York, New York
  - The Bronx, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Kettering, Ohio
  - Eugene, Oregon
  - Portland, Oregon
  - Springfield, Oregon
  - Tualatin, Oregon
  - Harrisburg, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Easley, South Carolina
  - Greenville, South Carolina
  - Spartanburg, South Carolina
  - Bartlett, Tennessee
  - Chattanooga, Tennessee
  - Germantown, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Southaven, Tennessee
  - Austin, Texas
  - Cedar Park, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Kyle, Texas
  - Round Rock, Texas
  - San Marcos, Texas
  - Salt Lake City, Utah
  - Arlington, Virginia
  - Fairfax, Virginia
  - Gainesville, Virginia
  - Leesburg, Virginia
  - Midlothian, Virginia
  - Richmond, Virginia
  - Winchester, Virginia
  - Woodbridge, Virginia
  - Seattle, Washington
  - Vancouver, Washington
  - Yakima, Washington
- Argentina (5):
  - Rosario, Santa Fe Province
  - Buenos Aires
  - Córdoba
  - San Miguel de Tucumán
  - Viedma
- Australia (7):
  - Greenslopes, Queensland
  - Camperdown
  - Kogarah
  - Perth
  - St Leonards
  - Wollongong
  - Woodville
- Austria (2):
  - Salzburg
  - Wels
- Belgium (3):
  - Brasschaat
  - Brussels
  - Duffel
- Brazil (8):
  - Salvador, Estado de Bahia
  - Rio de Janeiro, Rio de Janeiro
  - Passo Fundo, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Joinville, Santa Catarina
  - Ijuí
  - Porto Alegre
  - São Paulo
- Canada (11):
  - Edmonton, Alberta
  - Surrey, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - London, Ontario
  - Thunder Bay, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Montreal
  - Québec
  - Toronto
- Santiago, Chile
- Czechia (4):
  - Ostrava
  - Pardubice
  - Prague
  - Ústí nad Labem
- Denmark (3):
  - Herlev
  - Næstved
  - Odense
- France (14):
  - Besançon
  - Brest
  - Caen
  - Grenoble
  - Lille
  - Marseille
  - Paris
  - Pierre-Bénite
  - Rennes
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
  - Tours
  - Villejuif
- Germany (21):
  - Bad Berka
  - Berlin
  - Cologne
  - Erfurt
  - Essen
  - Esslingen am Neckar
  - Gauting
  - Großhansdorf
  - Halle
  - Hamburg
  - Hanover
  - Karlsruhe
  - Kassel
  - Leverkusen
  - Löwenstein
  - Mainz
  - Mannheim
  - München
  - Porta Westfalica
  - Rheine
  - Villingen-Schwenningen
- Hungary (5):
  - Deszk
  - Gyula
  - Mátraháza
  - Székesfehérvár
  - Szolnok
- Italy (25):
  - Ancona
  - Avellino
  - Aviano
  - Bari
  - Catania
  - Cremona
  - Cuneo
  - Florence
  - Livorno
  - Milan
  - Modena
  - Monza
  - Napoli
  - Novara
  - Orbassano
  - Padua
  - Palermo
  - Parma
  - Perugia
  - Roma
  - Rozzano
  - Sassari
  - Sondalo
  - Sora
  - Torino
- Mexico (5):
  - Mexico City, Mexico City
  - Monterrey, Nuevo León
  - Guadalajara
  - Mexico City
  - Oaxaca City
- Netherlands (3):
  - Enschede, ER
  - Helmond, HA
  - Amsterdam
- Peru (2):
  - Arequipa
  - Lima
- Poland (11):
  - Bystra
  - Krakow
  - Lublin
  - Olsztyn
  - Opole
  - Poznan
  - Prabuty
  - Rzeszów
  - Szczecin
  - Torun
  - Wałbrzych
- Romania (3):
  - Cluj-Napoca
  - Craiova
  - Oradea
- Russia (11):
  - Chelyabinsk
  - Irkutsk
  - Izhevsk
  - Kursk
  - Moscow
  - Novosibirsk
  - Pyatigorsk
  - Saint Petersburg
  - Tula
  - Tyumen
  - Veliky Novgorod
- Spain (16):
  - Barakaldo, Bilbao
  - Vigo, Pontevedra
  - A Coruña
  - Alicante
  - Barcelona
  - Madrid
  - Manresa
  - Málaga
  - Oviedo
  - Palma de Mallorca
  - Sabadell
  - San Cristóbal de La Laguna
  - Santiago de Compostela
  - Seville
  - Valencia
  - Zaragoza
- Sweden (2):
  - Linköping
  - Lund
- United Kingdom (7):
  - Guildford, Surrey
  - Aberdeen
  - Glasgow
  - London
  - Manchester
  - Nottingham
  - Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scagliotti G, von Pawel J, Novello S, Ramlau R, Favaretto A, Barlesi F, Akerley W, Orlov S, Santoro A, Spigel D, Hirsh V, Shepherd FA, Sequist LV, Sandler A, Ross JS, Wang Q, von Roemeling R, Shuster D, Schwartz B. Phase III Multinational, Randomized, Double-Blind, Placebo-Controlled Study of Tivantinib (ARQ 197) Plus Erlotinib Versus Erlotinib Alone in Previously Treated Patients With Locally Advanced or Metastatic Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2015 Aug 20;33(24):2667-74. doi: 10.1200/JCO.2014.60.7317. Epub 2015 Jul 13. PMID 26169611
- [Derived] Scagliotti GV, Novello S, Schiller JH, Hirsh V, Sequist LV, Soria JC, von Pawel J, Schwartz B, Von Roemeling R, Sandler AB. Rationale and design of MARQUEE: a phase III, randomized, double-blind study of tivantinib plus erlotinib versus placebo plus erlotinib in previously treated patients with locally advanced or metastatic, nonsquamous, non-small-cell lung cancer. Clin Lung Cancer. 2012 Sep;13(5):391-5. doi: 10.1016/j.cllc.2012.01.003. Epub 2012 Mar 21. PMID 22440336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1048 participants who met all inclusion criteria and no exclusion criteria were enrolled between 11 Jan 2011 and 18 Jul 2012 at 140 sites in Europe, 78 sites in United States, 32 sites in Latin America, and 20 sites in Canada/Australia. Of the 1048 participants, a total of 1037 participants received treatment.
Pre-assignment Details: Participants were to be randomized in a 1:1 ratio to tivantinib at 360 mg BID (total daily dose, 720 mg) + erlotinib at 150 mg QD, or placebo BID + erlotinib at 150 mg QD, to be administered in a double-blinded manner.
Groups:
- Tivantinib and Erlotinib: Participants who were randomized to receive Tivantinib 720 mg daily (360 mg twice a day) in combination with 150 mg of erlotinib, given once a day.
- Placebo and Erlotinib: Participants who were randomized to receive Tivantinib placebo given twice a day in combination with 150 mg of erlotinib, given once a day.
Period: Overall Study
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Started | 526 | 522
Did Not Receive Treatment | 6 | 5
Completed | 46 | 24
Not Completed | 480 | 498
Not completed — Progressive disease | 295 | 350
Not completed — Clinical disease progression | 54 | 36
Not completed — Adverse Event | 65 | 48
Not completed — Death | 22 | 29
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 1 | 2
Not completed — Withdrawal by Subject | 31 | 23
Not completed — 'Missing' or 'Terminated by sponsor' | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib | Total
Number analyzed (Participants) | 526 | 522 | 1048
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 320 | 326 | 646
  >=65 years | 206 | 196 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.10) | 61.1 (9.84) | 61.1 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 213 | 429
  Male | 310 | 309 | 619

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Following Treatment With Tivantinib (ARQ 197) Plus Erlotinib Compared to Placebo Plus Erlotinib in Previously Treated Participants With Locally Advanced or Metastatic, Non-Squamous, Non-Small-Cell Lung Cancer
Description: The overall survival (OS) was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Date of randomization up to date of death, up to approximately 1 year 11 months postdose
Population: Overall survival was assessed in the Intent-to-treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Number analyzed (Participants) | 526 | 522
months | 8.5 [7.1 to 9.3] | 7.8 [7.0 to 9.0]
Statistical Analysis 1: Comparison: Tivantinib and Erlotinib vs Placebo and Erlotinib; Test type: Superiority; p = 0.8086, Log Rank; Hazard Ratio (HR) = 0.981, 95% CI 2-sided [0.841 to 1.149] — Hazard ratio and the 95% confidence interval from stratified Cox-regression model (adjusting for number of prior therapies, gender, and smoking history)

2. Secondary Outcome: Progression-free Survival Following Treatment With Tivantinib (ARQ 197) Plus Erlotinib Compared to Placebo Plus Erlotinib in Previously Treated Participants With Locally Advanced or Metastatic, Non-Squamous, Non-Small-Cell Lung Cancer
Description: Progression-free Survival (PFS) was defined as the time from the date of randomization to the date of the first objective documentation of disease progression or date of death from any cause (whichever comes first). As per the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) criteria, progression was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Date of randomization to disease progression or death (whichever comes first), up to 1 year 11 months postdose
Population: Progression-free survival (PFS) was assessed in the Intent-to-treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Number analyzed (Participants) | 526 | 522
months | 3.6 [2.8 to 3.7] | 1.9 [1.9 to 2.0]

3. Secondary Outcome: Overall Survival in the Epidermal Growth Factor Receptor Gene Wild-Type Subpopulation Following Treatment With Tivantinib (ARQ 197) Plus Erlotinib Compared to Placebo Plus Erlotinib in Previously Treated Participants With Non-Squamous NSCLC
Description: The overall survival (OS) was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Date of randomization up to date of death, up to approximately 1 year 11 months postdose
Population: Overall survival was assessed in participants with the epidermal growth factor receptor wild-type gene.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Number analyzed (Participants) | 469 | 468
months | 7.2 [6.4 to 8.5] | 7.1 [6.3 to 7.8]

4. Secondary Outcome: Progression-free Survival in the Epidermal Growth Factor Receptor (EGFR) Gene Wild-Type Subpopulation Following Treatment With Tivantinib (ARQ 197) Plus Erlotinib Compared to Placebo Plus Erlotinib in Previously Treated Participants Non-Squamous NSCLC
Description: as for outcome 2
Time Frame: Date of randomization to disease progression or death (whichever comes first), up to 1 year 11 months postdose
Population: Progression-free survival (PFS) was assessed in participants with the epidermal growth factor receptor wild-type gene.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Number analyzed (Participants) | 469 | 468
months | 2.7 [1.9 to 3.6] | 1.9 [1.9 to 1.9]

5. Secondary Outcome: Best Overall Tumor Response Following Treatment With Tivantinib (ARQ 197) Plus Erlotinib Compared to Placebo Plus Erlotinib in Previously Treated Participants With Locally Advanced or Metastatic, Non-Squamous, Non-Small-Cell Lung Cancer
Description: The best overall response was defined as the best response (in the order of confirmed complete response [CR], confirmed partial response [PR], stable disease [SD], and progressive disease [PD]) among all overall responses recorded from the start of treatment until the participant withdrew from the study. If there was no tumor assessment after the first dose of study drug, the best overall response was classified as Inevaluable. Based on RECIST v1.1, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From baseline up to disease progression or the development of unacceptable toxicity (whichever occurs first), up to 1 year 11 months postdose
Population: Best overall response was assessed in the Intent-to-treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Number analyzed (Participants) | 526 | 522
Participants
  Complete response (CR) | 1 | 1
  Partial response (PR) | 53 | 33
  Objective response (CR+PR) | 54 | 34
  Stable disease (SD) | 187 | 133
  Progressive disease (PD) | 189 | 265
  Best response of SD or better | 241 | 167
  Inevaluable | 96 | 90

6. Secondary Outcome: Duration of Response Following Treatment With Tivantinib (ARQ 197) Plus Erlotinib Compared to Placebo Plus Erlotinib in Previously Treated Participants With Locally Advanced or Metastatic, Non-Squamous, Non-Small-Cell Lung Cancer
Description: Duration of response was defined for participants with confirmed CR or PR as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease. Duration of SD was defined for participants whose best response was SD as the time from the randomization date to the date of the first documentation of progressive disease.
Time Frame: From the date of first objective response (CR or PR) or SD to date of progressive disease, up to 1 year 11 months postdose
Population: Duration of response was assessed in the Intent-to-treat population.
Measure: Median (Full Range); unit: weeks
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Number analyzed (Participants) | 241 | 167
weeks
  Duration of objective response (CR or PR): number analyzed (Participants) | 54 | 34
  Duration of objective response (CR or PR) | 40.43 [0.1 to 56.1] | 47.86 [0.1 to 79.7]
  Duration of SD: number analyzed (Participants) | 187 | 133
  Duration of SD | 28.29 [7.9 to 80.0] | 23.86 [7.7 to 79.3]

7. Secondary Outcome: Treatment-Emergent Adverse Events Reported in ≥5% of Participants Following Treatment With Tivantinib (ARQ 197) Plus Erlotinib Compared to Placebo Plus Erlotinib in Previously Treated Participants With Non-Squamous, Non-Small-Cell Lung Cancer
Description: Treatment-emergent AEs (TEAEs) were defined as those AEs that occurred, having been absent before the study, or worsened in severity after the initiation of study treatment administration.
Time Frame: Baseline up to 30 days after last dose, up to 1 year 11 months postdose
Population: Adverse events were assessed in the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Number analyzed (Participants) | 520 | 517
Participants
  Any TEAE | 513 | 503
  Diarrhea | 180 | 212
  Rash | 172 | 193
  Decreased appetite | 151 | 149
  Dyspnea | 136 | 117
  Fatigue | 136 | 113
  Nausea | 121 | 123
  Cough | 110 | 91
  Asthenia | 100 | 90
  Dermatitis acneiform | 90 | 98
  Vomiting | 73 | 81
  Anemia | 83 | 51
  Weight decreased | 57 | 58
  Constipation | 57 | 54
  Pyrexia | 60 | 41
  Back pain | 54 | 47
  Dry skin | 41 | 56
  Pruritus | 31 | 44
  Neutropenia | 62 | 10
  Headache | 41 | 28
  Edema, peripheral | 37 | 29
  Insomnia | 33 | 29
  Abdominal pain | 34 | 27
  Noncardiac chest pain | 34 | 24
  Pneumonia | 35 | 22
  Dyspepsia | 30 | 24
  Abdominal pain, upper | 33 | 19
  Mucosal inflammation | 27 | 24
  Stomatitis | 22 | 27
  Hemoptysis | 30 | 19
  General physical health deterioration | 29 | 18
  Pain in extremity | 28 | 19
  Dizziness | 26 | 16
  Alopecia | 26 | 14

8. Secondary Outcome: Treatment-Emergent Adverse Events Related to Tivantinib/Placebo Experienced by ≥5% of Participants Following Treatment With Tivantinib (ARQ 197) Plus Erlotinib Compared to Placebo Plus Erlotinib in Previously Treated Participants With Non-Squamous NSCLC
Description: as for outcome 7
Time Frame: Baseline up to 30 days after last dose, up to 1 year 11 months postdose
Population: Adverse events were assessed in the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
Number analyzed (Participants) | 520 | 517
Participants
  TEAE related to tivantinib/placebo | 324 | 301
  Blood and Lymphatic System Disorders | 87 | 27
  Anemia | 44 | 17
  Neutropenia | 54 | 5
  Gastrointestinal Disorders | 165 | 163
  Diarrhea | 81 | 96
  Nausea | 63 | 68
  Vomiting | 31 | 39
  General Disorders & Administration Site Conditions | 135 | 114
  Asthenia | 43 | 38
  Fatigue | 78 | 63
  Metabolism and Nutrition Disorders | 82 | 84
  Decreased appetite | 73 | 71
  Skin and Subcutaneous Tissue Disorders | 148 | 130
  Dermatitis acneiform | 26 | 27
  Rash | 61 | 71

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline up to 30 days after last dose, up to approximately 1 year 11 months postdose.
Description: Treatment-emergent AEs (TEAEs) were defined as those AEs that occurred, having been absent before the study, or worsened in severity after the initiation of study treatment administration. Safety events were assessed in the Safety Population.
Arm/Group | Tivantinib and Erlotinib | Placebo and Erlotinib
All-Cause Mortality (participants affected / at risk) | 77/520 | 65/517
Serious Adverse Events (participants affected / at risk) | 219/520 | 191/517
Other Adverse Events (participants affected / at risk) | 513/520 | 503/517
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tivantinib and Erlotinib (N=520) | Placebo and Erlotinib (N=517)
Anemia (Blood and lymphatic system disorders) | 16 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 15 | 2
Neutropenia (Blood and lymphatic system disorders) | 11 | 1
General physical health deterioration (General disorders) | 15 | 13
Pneumonia (Infections and infestations) | 20 | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 29 | 25
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 18
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 3 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Pericarditis restrictive (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 6
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 2
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 6
Oesophageal disorder (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4
Asthenia (General disorders) | 3 | 5
Fatigue (General disorders) | 4 | 2
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multi-organ disorder (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 3 | 0
Performance status decreased (General disorders) | 5 | 3
Pyrexia (General disorders) | 1 | 5
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 5
Bronchopneumonia (Infections and infestations) | 3 | 2
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Genital infection (Infections and infestations) | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 4
Perirectal abscess (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 3
Sepsis (Infections and infestations) | 5 | 2
Septic shock (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3
Wound infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Stemal fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Coagulation test abnormal (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 0 | 2
Hepatic enzyme increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 0
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 2 | 0
White blood cell count increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Aphasia (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Brain compression (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 4
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 5
Demyelination (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 2 | 0
Epiduritis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 2 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2
Nervous system disorder (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 2
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diffuse aveolar damage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 2
Embolism arterial (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Superior vena caval occulsion (Vascular disorders) | 0 | 3
Venous insufficiency (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tivantinib and Erlotinib (N=520) | Placebo and Erlotinib (N=517)
Anaemia (Blood and lymphatic system disorders) | 83 | 51
Neutropenia (Blood and lymphatic system disorders) | 62 | 10
Abdominal pain (Gastrointestinal disorders) | 34 | 27
Abdominal pain, upper (Gastrointestinal disorders) | 33 | 19
Constipation (Gastrointestinal disorders) | 57 | 54
Diarrhea (Gastrointestinal disorders) | 180 | 212
Dyspepsia (Gastrointestinal disorders) | 30 | 24
Nausea (Gastrointestinal disorders) | 121 | 123
Stomatitis (Gastrointestinal disorders) | 22 | 27
Vomiting (Gastrointestinal disorders) | 73 | 81
Asthenia (General disorders) | 100 | 90
Fatigue (General disorders) | 136 | 113
General physical health deterioration (General disorders) | 29 | 18
Mucosal inflammation (General disorders) | 27 | 24
Noncardiac chest pain (General disorders) | 34 | 24
Edema, peripheral (General disorders) | 37 | 29
Pyrexia (General disorders) | 60 | 41
Pneumonia (Infections and infestations) | 35 | 22
Weight decreased (Investigations) | 57 | 58
Decreased appetite (Metabolism and nutrition disorders) | 151 | 149
Back pain (Musculoskeletal and connective tissue disorders) | 54 | 47
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 19
Dizziness (Nervous system disorders) | 26 | 16
Headache (Nervous system disorders) | 41 | 28
Insomnia (Psychiatric disorders) | 33 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 110 | 91
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 136 | 117
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 30 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 14
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 90 | 98
Dry skin (Skin and subcutaneous tissue disorders) | 41 | 56
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 44
Rash (Skin and subcutaneous tissue disorders) | 172 | 193

LIMITATIONS AND CAVEATS:
Based on the interim OS data, the study was terminated due to the protocol-defined stopping boundary for futility being met. The study would not meet its primary endpoint of improved OS in the ITT population. There were no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No